CLINICAL TRIAL: NCT02656173
Title: A Phase 4, Double-blind, Randomized, Placebo-controlled Multicenter Study to Evaluate the Efficacy and Safety of Mirabegron in Japanese and Korean Male Patients With Overactive Bladder Under Treatment With the α-Blocker Tamsulosin for Benign Prostatic Hyperplasia
Brief Title: A Phase 4 Study to Evaluate the Efficacy, Safety, and Tolerability of Mirabegron in Male Subjects With Overactive Bladder (OAB) Symptoms, While Taking the Alpha Blocker for Benign Prostatic Hypertrophy (BPH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-MA-3016
Record Dates: First submitted 2016-01-13; First posted 2016-01-14 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder
Keywords: Tamsulosin; Overactive bladder; Benign prostatic hypertrophy; Mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — mirabegron; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mirabegron 50 mg (Experimental): Participants who received mirabegron 50 mg once a day along with tamsulosin 0.2 mg for 12 weeks
  Interventions: Drug: Mirabegron; Drug: Tamsulosin
- Placebo (Experimental): Participants who received matching placebo once a day along with tamsulosin 0.2 mg for 12 weeks.
  Interventions: Drug: Placebo; Drug: Tamsulosin

INTERVENTIONS:
Drug: Mirabegron — Oral tablet
  Other Names: YM178
  Arms: Mirabegron 50 mg
Drug: Placebo — Oral tablet
  Arms: Placebo
Drug: Tamsulosin — Oral tablet

SUMMARY:
The primary objective of the study was to investigate the efficacy of mirabegron versus placebo in male patients with OAB symptoms while taking the alpha blocker, tamsulosin, for BPH.

ELIGIBILITY:
Inclusion Criteria:

at Visit 1 (Screening):

* Patient had been under treatment with tamsulosin 0.2mg for at least 4 weeks before the start of the Screening period.
* Patient with a history of an average of at least 2 episodes of urgency per 24 hours and an average of 8 or more micturitions per 24 hours during the last 3 days before the start of the Screening period (verified by interview).
* Patient who had no wish to have children in the future (Unique to Japan).
* Male subjects and their female spouses/partners who were of childbearing potential must be using highly effective contraception consisting of two forms of birth control (at least one of which must be a barrier method), starting at Screening, continuing throughout the study period, and for 28 days after the final study drug administration.
* Subject must not donate sperm, starting at Screening, continuing throughout the study period, and for 28 days after the final study drug administration.
* Patient was willing and able to complete the micturition diary and questionnaires correctly.
* Subject agreed not to participate in another interventional study while receiving treatment in this study.

at Visit 2 (Baseline):

* Subject with an average of at least 2 episodes of urgency per 24 hours and an average of 8 or more micturitions per 24 hours based on a 3-day micturition diary from the Screening period.

Exclusion Criteria:

at Visit 1 (Screening):

* Patient with suspected symptoms of OAB, with onset only transient (e.g., drug-induced, psychogenic).
* Patient with PVR urine volume >100 mL or Q max <5 mL/sec.
* Patient with prostate-specific antigen (PSA) ≥4 ng/mL.
* Patient with neurogenic bladder (e.g., spinal-cord lesions or other damage that will clearly affect urination; multiple sclerosis; Parkinson's disease) or a history of surgery that caused damage to the pelvic plexus.
* Patient with urethral stricture or bladder-neck stenosis.
* Patient with diabetic neuropathy complications.
* Patient who had undergone a surgical procedure, previous pelvic radiation therapy, or hyperthermia therapy that may affect urinary tract function.
* Patient with significant stress incontinence or postsurgical prostate incontinence, as determined by the Investigator.
* Patient with an indwelling catheter or practices intermittent self-catheterization.
* Patient with 3 or more episodes of recurrent urinary tract infection (UTI) within the last 6 months.
* Patient with a UTI; prostatitis; chronic inflammation, such as interstitial cystitis; urinary calculus; or previous or current malignant disease of the pelvic organs.
* Patient with a concurrent malignancy or history of any malignancy (within the past 5 years), except for non-metastatic basal-cell or squamous-cell carcinoma of the skin that had been treated successfully.
* Patient with serious heart disease, liver disease, kidney disease, immunological disease, lung disease.
* Patient who had received intravesical injection within the last 12 months with botulinum toxin, resiniferatoxin, or capsaicin.
* Patient who had received electrostimulation therapy for OAB.
* Patient who had received a bladder training program or pelvic floor exercises <28 days prior to the start of the Screening period.
* Patient with postural hypotension or syncope, hypokalemia, or closed-angle glaucoma.
* Patient with evidence of QT prolongation on electrocardiogram (ECG), defined as QTcF >450 msec.
* Patient with severe uncontrolled hypertension, defined as sitting systolic blood pressure (SBP) >180 mmHg and/or diastolic blood pressure (DBP) >110 mmHg.
* Patient with a clinically significant ECG abnormality, as determined by the Investigator.
* Patient who had severe renal impairment, defined as an estimated glomerular filtration rate of <29 mL/min/1.73m2; end-stage renal disease; or is undergoing dialysis.
* Patient with aspartate transaminase (AST) or alanine transaminase (ALT) >2 times the upper limit of normal (ULN), or gamma-glutamyl transferase (γ-GT) >3 times the ULN and considered clinically significant by the Investigator.
* Patient with moderate or severe hepatic impairment, defined as Child-Pugh Class B or C.
* Patient with hypersensitivity to any of the components of mirabegron, other beta-adrenergic receptor (β-AR) agonists, or any of the inactive ingredients.
* Patient with ongoing alcohol and/or drug abuse.
* Patient with or a history of mood disorder, neurotic disorder, or schizophrenia.
* Patient with dementia, cognitive dysfunction, or clinically significant cerebrovascular disorder.
* Patient who had been treated with an experimental device <84 days or received an investigational agent <84 days prior to the start of the Screening period.
* Patient had used any prohibited concomitant medication <28 days (but, <1 year for 5α-reductase inhibitors) before the start of the Screening period.
* Patient with any clinically significant condition, which in the opinion of the Investigator, made the subject unsuitable for study participation.
* Patient who was involved in the conduct of the study as an employee of the Astellas group, a third party associated with the study, or the study site team.

at Visit 2 (Baseline):

* Subject fulfills any exclusion criteria of Visit 1 at Visit 2.
* Subject was noncompliant during the 4 week tamsulosin Screening period, defined as taking less than 80% or greater than 120% of prescribed dose of study medication.
* Subject had an average total daily urine volume >3000 mL, as recorded in the 3-day micturition diary.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (58):
- Japan (53):
  - Site JP81046, Aichi
  - Site JP81009, Chiba
  - Site JP81045, Chiba
  - Site JP81041, Fukuoka
  - Site JP81042, Fukuoka
  - Site JP81043, Fukuoka
  - Site JP81044, Fukuoka
  - Site JP81048, Fukuoka
  - Site JP81004, Gunma
  - Site JP81005, Gunma
  - Site JP81001, Hokkaido
  - Site JP81002, Hokkaido
  - Site JP81003, Hokkaido
  - Site JP81038, Hyōgo
  - Site JP81039, Hyōgo
  - Site JP81040, Hyōgo
  - Site JP81024, Kanagawa
  - Site JP81056, Kanagawa
  - Site JP81051, Kochi
  - Site JP81052, Kochi
  - Site JP81047, Kumamoto
  - Site JP81025, Osaka
  - Site JP81026, Osaka
  - Site JP81027, Osaka
  - Site JP81028, Osaka
  - Site JP81029, Osaka
  - Site JP81030, Osaka
  - Site JP81031, Osaka
  - Site JP81032, Osaka
  - Site JP81033, Osaka
  - Site JP81034, Osaka
  - Site JP81035, Osaka
  - Site JP81036, Osaka
  - Site JP81037, Osaka
  - Site JP81053, Osaka
  - Site JP81054, Osaka
  - Site JP81006, Saitama
  - Site JP81007, Saitama
  - Site JP81008, Saitama
  - Site JP81050, Shizuoka
  - Site JP81010, Tokyo
  - Site JP81011, Tokyo
  - Site JP81012, Tokyo
  - Site JP81013, Tokyo
  - Site JP81014, Tokyo
  - Site JP81015, Tokyo
  - Site JP81016, Tokyo
  - Site JP81017, Tokyo
  - Site JP81018, Tokyo
  - Site JP81019, Tokyo
  - Site JP81020, Tokyo
  - Site JP81021, Tokyo
  - Site JP81022, Tokyo
- South Korea (5):
  - Site KR00001, Seoul
  - Site KR00002, Seoul
  - Site KR00003, Seoul
  - Site KR00004, Seoul
  - Site KR00005, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kakizaki H, Lee KS, Katou D, Yamamoto O, Sumarsono B, Uno S, Yamaguchi O. Mirabegron Add-On Therapy to Tamsulosin in Men with Overactive Bladder: Post Hoc Analyses of Efficacy from the MATCH Study. Adv Ther. 2021 Jan;38(1):739-757. doi: 10.1007/s12325-020-01517-5. Epub 2020 Nov 27. PMID 33245533
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male participants with overactive bladder (OAB) under treatment with the α-blocker tamsulosin for benign prostatic hyperplasia (BPH) were enrolled in Japan (53 sites) and Korea (5 sites).
Pre-assignment Details: Eligible participants received tamsulosin 0.2 mg and placebo orally once a day after breakfast for 4 weeks. Subsequently, participants who met the eligibility criteria at the end of this 4 week screening period were randomized 1:1 to mirabegron 50 mg group or placebo group with tamsulosin 0.2 mg orally once a day after breakfast for 12 weeks.
Groups:
- Placebo: Participants received matching placebo once a day along with tamsulosin 0.2 mg for 12 weeks.
- Mirabegron 50mg: Participants received mirabegron 50 mg once a day along with tamsulosin 0.2 mg for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Mirabegron 50mg
Started | 285 | 283
Received Treatment | 284 | 282
Completed | 272 | 272
Not Completed | 13 | 11
Not completed — Deviation from the Eligible Criteria | 3 | 2
Not completed — Adverse Event | 7 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Miscellaneous | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirabegron 50mg | Total
Number analyzed (Participants) | 285 | 283 | 568
Age, Continuous [Mean (Standard Deviation); unit: year] | 65.6 (9.0) | 65.3 (8.5) | 65.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 285 | 283 | 568
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 285 | 283 | 568
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 269 | 269 | 538
  Korean | 16 | 14 | 30
Mean number of micturitions per 24 hours [Mean (Standard Deviation); unit: micturitions] — A micturition was defined as any voluntary micturition (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by participants on a 3-day micturition diary before each visit. Population: Full analysis set (FAS) consisted of all participants who were randomized and received ≥ 1 dose of double-blind study drug and had a baseline micturition measurement and ≥ 1 post-baseline micturition measurement.
  micturitions
    number analyzed (Participants) | 283 | 282 | 565
    (all) | 10.760 (2.355) | 10.401 (2.236) | 10.581 (2.301)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment (EoT) in Mean Number of Micturitions Per 24 Hours
Description: A micturition was defined as any voluntary micturition (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated from data recorded by participants on a 3-day micturition diary before each visit.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: Full analysis set (FAS) consisted of all subjects who were randomized and received ≥ 1 dose of double-blind study drug and had a baseline micturition measurement and ≥ 1 post-baseline micturition measurement. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: micturitions
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 280 | 278
micturitions | -0.90 (1.91) | -1.35 (1.81)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; Analysis of Covariance (ANCOVA) was used for analysis, including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p < 0.001, ANCOVA; least square mean difference = -0.52, 95% CI 2-sided [-0.82 to -0.21]

2. Primary Outcome: Change From Baseline to Weeks 4, 8, 12 in Mean Number of Micturitions Per 24 Hours
Description: as for outcome 1
Time Frame: Baseline and week 4, 8 and 12
Population: FAS.
Measure: Mean (Standard Deviation); unit: micturitions
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 283 | 282
micturitions
  Week 4: number analyzed (Participants) | 279 | 278
  Week 4 | -0.08 (1.66) | -0.55 (1.45)
  Week 8: number analyzed (Participants) | 274 | 275
  Week 8 | -0.36 (1.87) | -0.76 (1.83)
  Week 12: number analyzed (Participants) | 271 | 272
  Week 12 | -0.92 (1.90) | -1.36 (1.83)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; Mixed Model Repeated Measure (MMRM) was used for analysis, which included the baseline as a covariate, treatment group, analysis visits and region as a fixed effect, subject as random effect and including interaction of [treatment group x visit] for FAS; Test type: Superiority; p < 0.001, mixed model repeated measure; least square mean difference = -0.48, 95% CI 2-sided [-0.78 to -0.17]

3. Secondary Outcome: Change From Baseline to EoT in Mean Number of Urgency Episodes Per 24 Hours
Description: An urgency episode was defined as a complaint of a sudden, compelling desire to pass urine, which is difficult to defer. The mean number of urgency episodes per 24 hours was calculated from data recorded by participants on a 3-day micturition diary before each visit.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS who had at least 1 urgency episode at baseline. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: urgency episodes
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 280 | 278
urgency episodes | -1.66 (2.48) | -1.89 (2.00)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; Analysis of Covariance (ANCOVA) was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.112, ANCOVA; least square mean difference = -0.28, 95% CI 2-sided [-0.63 to 0.07]

4. Secondary Outcome: Change From Baseline to EoT in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: An urgency incontinence episode was defined as any episode when both urgency and incontinence occurred concurrently. The mean number of urgency incontinence episodes per 24 hours was calculated from data recorded by participants on a 3-day micturition diary before each visit.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS who had at least 1 urgency incontinence episode at baseline. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: urgency incontinence episodes
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 74 | 86
urgency incontinence episodes | -0.65 (1.31) | -0.75 (0.80)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; Stratified Rank Analysis of Covariance (RANCOVA), including the rank score for change from Baseline to End of Treatment stratified by region as the dependent variable, treatment group and region as fixed factors and the rank score for baseline stratified by region as a covariate for FAS; Test type: Superiority; p = 0.186, Stratified Rank Analysis of Covariance; Cochran-Mantel-Haenszel Statistics = 1.75

5. Secondary Outcome: Change From Baseline to EoT in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as the complaint of any involuntary leakage of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by participants on a 3-day micturition diary before each visit.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS who had at least 1 incontinence episode at baseline. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: incontinence episodes
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 80 | 89
incontinence episodes | -0.72 (1.30) | -0.77 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.760, Stratified Rank Analysis of Covariance; Cochran-Mantel-Haenszel Statistics = 0.09

6. Secondary Outcome: Change From Baseline to EoT in Mean Number of Nocturia Episodes
Description: A nocturia episode was defined as a micturition episode initiated between night time. Night time was defined as the period between sleep onset time and the wake-up time the following day (micturitions at the same time as the wake-up time were excluded). The mean number of nocturia episodes per 24 hours was calculated from data recorded by participants on a 3-day micturition diary before each visit.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS who had at least 1 nocturia episode at baseline. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: nocturia episodes
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 255 | 245
nocturia episodes | -0.35 (0.86) | -0.31 (0.95)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.646, ANCOVA; Least square mean difference = -0.03, 95% CI 2-sided [-0.18 to 0.11]

7. Secondary Outcome: Change From Baseline to EoT in Mean Volume Voided Per Micturition
Description: The mean volume voided per micturition was calculated from data recorded by participants on a 3-day micturition diary before each visit.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS who had volume voided as > 0. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 272 | 272
mL | 2.632 (32.959) | 14.995 (35.486)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = 12.08, 95% CI 2-sided [6.33 to 17.84]

8. Secondary Outcome: Change From Baseline to EoT in Total Overactive Bladder Symptom Score (OABSS)
Description: The OABSS is a 4-item questionnaire that assesses urinary frequency. Total score was the sum total of the score of each item (ranges: 0-15). Negative change means improvement.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: FAS. EoT value was defined as last post-baseline assessment during the double-blind study period for which the efficacy data are available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 283 | 281
units on a scale | -2.2 (2.4) | -2.8 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.001, ANCOVA; Least square mean difference = -0.65, 95% CI 2-sided [-1.04 to -0.26]

9. Secondary Outcome: Change From Baseline to EoT in OABSS Subscale Scores
Description: Each OABSS subscale score was based on each question in the questionnaire: Daytime Frequency ("How many times do you typically urinate from waking in the morning until sleeping at night?" where scores range from 0-2), Nighttime Frequency ("How many times do you typically wake up to urinate from sleeping at night until waking in the morning?" where scores range from 0-3), Urgency ("How often do you have a sudden desire to urinate, which is difficult to defer?" where scores range from 0-5), Urgency Incontinence ("How often do you leak urine because you cannot defer the sudden desire to urinate?" where scores range from 0-5). A higher score is indicative of worse condition and a negative change from baseline indicates an improvement.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 283 | 281
units on a scale
  Daytime Frequency | -0.2 (0.5) | -0.3 (0.5)
  Nighttime Frequency | -0.2 (0.7) | -0.3 (0.8)
  Urgency | -1.3 (1.5) | -1.5 (1.4)
  Urgency Incontinence | -0.4 (1.1) | -0.7 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; Subscale: Daytime Frequency. Analysis of Covariance (ANCOVA) was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.006, ANCOVA; Least square mean difference = -0.11, 95% CI 2-sided [-0.19 to -0.03]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50mg; Subscale: Nighttime Frequency. ANCOVA was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.174, ANCOVA; Least square mean difference = -0.08, 95% CI 2-sided [-0.19 to 0.03]
Statistical Analysis 3: Comparison: Placebo vs Mirabegron 50mg; Subscale: Urgency. ANCOVA was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.037, ANCOVA; Least square mean difference = -0.26, 95% CI 2-sided [-0.50 to -0.02]
Statistical Analysis 4: Comparison: Placebo vs Mirabegron 50mg; Subscale: Urgency Incontinence. ANCOVA was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.014, ANCOVA; Least square mean difference = -0.18, 95% CI 2-sided [-0.32 to -0.04]

10. Secondary Outcome: Change From Baseline to EoT in Total International Prostate Symptom Score (IPSS)
Description: The IPSS included an 7-item questionnaire that assesses urinary frequency and incomplete voiding along with a QoL assessment. Total IPSS score was the sum total of the score (range: 0-35) of each item (Questions 1-7). Negative change means improvement.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 283 | 281
units on a scale | -3.4 (5.0) | -4.4 (4.7)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Least square mean difference = -1.19, 95% CI 2-sided [-1.94 to -0.44]

11. Secondary Outcome: Change From Baseline to EoT in IPSS Subscale Scores
Description: IPSS subscale scores was calculated by following each formula. Storage subscale was derived as sum of scores for questions 2, 4, and 7 (range: 1-15). Voiding subscale-1 was derived as sum of scores for questions 3, 5, and 6 (range: 1-15). Voiding subscale-2 was derived as sum of voiding subscale-1 and the score for question 1 (range: 1-20). Individual scores and IPSS Quality of Life (QoL) score was the score of each item (range: 1-6) (Questions 1-7 and QoL item). A higher score is indicative of worse condition and a negative change from baseline indicates an improvement.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 283 | 281
units on a scale
  Storage Subscale | -1.7 (2.4) | -2.4 (2.2)
  Voiding Subscale-1 | -1.3 (2.8) | -1.4 (2.9)
  Voiding Subscale-2 | -1.7 (3.4) | -2.0 (3.4)
  Quality of Life Item | -0.9 (1.3) | -1.2 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; Subscale: Storage Subscale. Analysis of Covariance (ANCOVA) was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -0.78, 95% CI 2-sided [-1.13 to -0.43]
Statistical Analysis 2: Comparison: Placebo vs Mirabegron 50mg; Subscale: Voiding Subscale-1. ANCOVA was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.167, ANCOVA; Least square mean difference = -0.30, 95% CI 2-sided [-0.72 to 0.13]
Statistical Analysis 3: Comparison: Placebo vs Mirabegron 50mg; Subscale: Voiding Subscale-2. ANCOVA was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.103, ANCOVA; Least square mean difference = -0.42, 95% CI 2-sided [-0.93 to 0.09]
Statistical Analysis 4: Comparison: Placebo vs Mirabegron 50mg; Subscale: Quality of Life (QoL) Item. ANCOVA was used for analysis including treatment group and region as fixed factors and baseline as a covariate; Test type: Superiority; p = 0.009, ANCOVA; Least square mean difference = -0.29, 95% CI 2-sided [-0.51 to -0.07]

12. Secondary Outcome: Change From Baseline to EoT in Symptom Bother as Assessed by the Overactive Bladder Questionnaire (OAB-q)
Description: The OAB-q was a 33-item questionnaire, which consisted of an 8-item symptom bother scale and 25 health-related QoL items that form 4 subscales (coping, concern, sleep, and social interaction) and a total health-related QoL score.
  Symptom Bother was derived as sum of scores for questions 1-8 (range: 0-100). Higher Symptom Bother is indicative of greater symptom bother.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 280 | 279
units on a scale | -11.53 (17.06) | -16.09 (15.99)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = -4.52, 95% CI 2-sided [-6.91 to -2.13]

13. Secondary Outcome: Change From Baseline to EoT in Total Health-Related QoL (HRQoL) Scores as Assessed by the OAB-q
Description: The OAB-q was a 33-item questionnaire, which consisted of an 8-item symptom bother scale and 25 health-related QoL items that form 4 subscales (coping, concern, sleep, and social interaction) and a total health-related QoL score.
  Total HRQL score was derived as sum of HRQL subscale scores (range: 25-150). Higher total HRQL score is indicative of better HRQL.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 280 | 279
units on a scale | 6.54 (11.98) | 9.70 (12.04)
Statistical Analysis 1: Comparison: Placebo vs Mirabegron 50mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Least square mean difference = 2.79, 95% CI 2-sided [1.13 to 4.44]

14. Secondary Outcome: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events (TEAE) was defined as an adverse event (AE) with onset during the double-blind treatment period or an AE with onset during the screening period with worsening severity during the double-blind treatment period. The investigator assessed the severity of AEs as follows: Mild: No disruption of normal daily activities; Moderate: Affected normal daily activities; Severe: Inability to perform daily activities. A drug-related TEAE was a TEAE with at least a possible relationship to the study drug as assessed by the investigator. Serious TEAE was an AE considered serious.
Time Frame: From first dose of study drug up to Week 12
Population: Safety Analysis Set (SAF) consisted of all participants who received at least 1 dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 284 | 282
Participants
  Any TEAEs | 64 | 66
  Mild | 57 | 56
  Moderate | 6 | 8
  Severe | 1 | 2
  Drug-related TEAEs | 18 | 11
  TEAEs leading to death | 0 | 0
  Serious TEAEs | 3 | 6
  Drug-related serious TEAEs | 1 | 0
  TEAEs leading to discontinuation of study drug | 4 | 4
  Drug-related TEAEs leading to disc. of study drug | 3 | 0

15. Secondary Outcome: Change From Baseline to EoT in Postvoid Residual (PVR) Volume
Description: PVR was measured by ultrasonography.
Time Frame: Baseline and EoT (up to 12 weeks)
Population: SAF. EoT value was defined as last post-baseline assessment during the double-blind study period for which the safety data are available.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 283 | 281
mL | -0.97 (21.42) | 2.72 (24.94)

16. Secondary Outcome: Change From Baseline to EoT in Maximum Urine Flow Rate (Qmax)
Description: Urine flow rate was volume voided per micturition (voided volume) divided by time for the micturition (flow time).
Time Frame: Baseline and EoT (up to 12 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Placebo: Patients received matching placebo once a day along with tamsulosin 0.2 mg for 12 weeks.
- Mirabegron 50mg: Patients received mirabegron 50 mg once a day along with tamsulosin 0.2 mg for 12 weeks.
Arm/Group | Placebo | Mirabegron 50mg
Number analyzed (Participants) | 280 | 278
mL | 0.20 (5.70) | -0.25 (5.82)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 12
Description: Safety Anlysis Set (SAF). The SAF consisted of participants who received at least 1 dose of the study drug for the treatment period.
Arm/Group | Placebo | Mirabegron 50mg
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/282
Serious Adverse Events (participants affected / at risk) | 3/284 | 6/282
Other Adverse Events (participants affected / at risk) | 17/284 | 18/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=284) | Mirabegron 50mg (N=282)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=284) | Mirabegron 50mg (N=282)
Nasopharyngitis (Infections and infestations) | 17 (21) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT02656173/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02656173/SAP_000.pdf